CLINICAL TRIAL: NCT02949466
Title: Additional Therapeutic Effects of Triamcinolone to Hyaluronic Acid on Knee Osteoarthritis: A Double Blind, Randomized-controlled Clinical Trial
Brief Title: Additional Effects of Triamcinolone to Hyaluronic Acid on Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST 105-2314-B-341-002
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Physical Activity; Functional Performance
Keywords: knee osteoarthritis; triamcinolone; therapeutic effects
MeSH Terms: conditions — Motor Activity; Osteoarthritis, Knee | interventions — Triamcinolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triamcinolone and hyaluronic acid group (Experimental): combined triamcinolone (Triamcinolone 10 mg 1cc) and hyaluronic acid (2 cc) injections: one injection per week, for 3 weeks, to compare the additional therapeutic effects of combined triamcinolone and hyaluronic acid injections to hyaluronic acid injections
  Interventions: Drug: Triamcinolone; Device: Hyaluronic acid
- hyaluronic acid group (Active Comparator): hyaluronic acid (2cc) injection: one injection per week, for 3 weeks, to compare the additional therapeutic effects of combined triamcinolone and hyaluronic acid injections to hyaluronic acid injections
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Drug: Triamcinolone — compare the additional therapeutic effects of triamcinolone combined with hyaluronic acid injections to hyaluronic acid injections only to patients with knee osteoarthritis
  Other Names: corticosteroids
  Arms: triamcinolone and hyaluronic acid group
Device: Hyaluronic acid — compare the additional therapeutic effects of triamcinolone combined with hyaluronic acid injections to hyaluronic acid injections only to patients with knee osteoarthritis

SUMMARY:
Using a double-blind, randomized controlled design to investigate the additional therapeutic effects of 3 times of combined triamcinolone and hyaluronic acid injections to 3 times of hyaluronic acid injections to patients with knee osteoarthritis.

DETAILED DESCRIPTION:
A total of 56 patients will be enrolled and randomized into two groups, including 3 times of triamcinolone combined hyaluronic acid injections group and 3 times of hyaluronic acid injections group.

The triamcinolone combined hyaluronic acid injections group will receive 3 times of triamcinolone combined hyaluronic acid injection per week in three weeks; the hyaluronic acid group will receive hyaluronic acid injection in three weeks.

Physical activities and functional performance will be evaluated at before injection, at after one week, one month, three months, and six months of completion of 3 times of injections.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis with Kellgren/Lawrence grade II or III

Exclusion Criteria:

* who have neurological deficit, such as stroke who have implant in knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Functional performance assessed with the Western Ontario and McMaster Universities Osteoarthritis Index | changes from baseline to at after one week, one month, three months, and six months of completion of injections
  Western Ontario and McMaster Universities Osteoarthritis Index

SECONDARY OUTCOMES:
10 meter walk test | changes from baseline to at after one week, one month, three months, and six months of completion of injections
  10 meter walk as fast as possible
Quality of life assessed with the Knee Injury and Osteoarthritis Outcome Score | changes from baseline to at after one week, one month, three months, and six months of completion of injections
  Knee Injury and Osteoarthritis Outcome Score
5 times rapid chair rising test | changes from baseline to at after one week, one month, three months, and six months of completion of injections
  rapid chair rising for 5 times as fast as possible

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CP, Lee WC, Hsieh RL. Effects of Repeated Co-Injections of Corticosteroids and Hyaluronic Acid on Knee Osteoarthritis: A Prospective, Double-Blind Randomized Controlled Trial. Am J Med. 2022 May;135(5):641-649. doi: 10.1016/j.amjmed.2021.11.016. Epub 2021 Dec 24. PMID 34958762